CLINICAL TRIAL: NCT05853263
Title: Pediatric Analgesia After Cardiac Surgery; Morphine IV Versus Paracetamol IV After Cardiac Surgery in Neonates and Infants.
Brief Title: Morphine IV vs Paracetamol IV in Neonates and Infants After Cardiac Surgery
Acronym: PACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: KU Leuven (Other); UMC Utrecht (Other); University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Gerdien (G.A.) Zeilmaker-Roest, clinical investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL 53085.078.15
Record Dates: First submitted 2023-03-25; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Analgesia; Congenital Heart Disease; Surgery
Keywords: morphine; paracetamol; neonates; infants; child; analgesia; congenital heart defect; cardiopulmonary bypass; congenital cardiac surgery; pharmacokinetics
MeSH Terms: conditions — Agnosia; Heart Defects, Congenital | interventions — Acetaminophen; Morphine

STUDY DESIGN:
Intervention Model Description: prospective, double blind, randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind, randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- morphine (Other): Standard care, continuous morphine IV.
  Interventions: Drug: Morphine
- paracetamol (Active Comparator): intervention group, intermittent paracetamol IV
  Interventions: Drug: paracetamol

INTERVENTIONS:
Drug: paracetamol — paracetamol IV to substitute morphine IV.
  Other Names: Acetominophen
  Arms: paracetamol
Drug: Morphine — standard care
  Arms: morphine

SUMMARY:
The goal of this clinical trial is to compare pain management in neonates and infants under 3 years of age undergoing cardiac surgery with use of cardiopulmonary bypass. Patients will be randomized to either continuous morphine IV (standard) of intermittent paracetamol IV (intervention).

The investigators' hypothesis is that intermittent IV paracetamol is effective as the primary analgesic drug in post-cardiac surgery patients up to 3 years of age and that the use of IV paracetamol will reduce overall morphine requirements.

DETAILED DESCRIPTION:
Congenital heart disease accounts for almost one third of all congenital anomalies. Surgical intervention is necessary in 55% within the first year of life and in 67% during the first three years of life.

Morphine is the drug of first choice worldwide for pain relief after major surgery in neonates and children. However, morphine can cause unwanted hemodynamic and respiratory reactions and therefore patients could potentially benefit from a non-opioid analgesic.

In a recent randomized controlled trial, intravenous (IV) paracetamol was compared with morphine as a primary analgesic drug in non-cardiac post-operative children up to 1 year. IV paracetamol was equally effective in pain relief, and no difference in rescue analgesics was shown between groups. The IV paracetamol group had a lower cumulative morphine dose the first 48 h after surgery and less adverse drug reactions.

Whether these results also apply to neonates and children after cardiac surgery is unclear. Pharmacokinetic (PK) parameters are assumed to be different in patients during and after cardiac surgery compared with non-cardiac surgery due to use of the cardiopulmonary bypass (CPB).

Hypothesis The investigators' hypothesis is that intermittent IV paracetamol is effective as the primary analgesic drug in post-cardiac surgery patients up to 3 years of age and that the use of IV paracetamol will reduce overall morphine requirements.

This hypothesis is currently being tested at three level-4 PICUs in the Netherlands and Belgium (Erasmus MC-Sophia Rotterdam, Wilhelmina Children's Hospital University Medical Center (UMC) Utrecht, Beatrix Children's Hospital UMC Groningen, University Hospital (UZ) Leuven).

All participants will receive a loading dose of morphine after cardiac surgery. After this, participants will be randomized to either standard care (morphine continuous IV) or intervention group (intermittent paracetamol IV).

Validated pain and sedations assessment tools will be used to adjust pain treatment if necessary. Rescue morphine as available for both groups.

A double blind study design is used, with a dummy saline continuous infusion in the paracetamol group and a dummy saline intermittent infusion in de continuous morphine group.

Study medication is stopped 48 hours after surgery and patients are transferred to open label morphine and paracetamol when applicable.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Neonates/infants who are 0-36 months old
* Cardiac surgery with the use of CPB.

Exclusion Criteria:

* No informed consent
* Known allergy to or intolerance of paracetamol or morphine
* Administration of opioids in the 24 h prior to surgery
* Hepatic dysfunction defined as three times the reference value of alanine aminotransferase/aspartate aminotransferase (ALAT/ASAT)
* Renal insufficiency at least RIFLE category Risk prior to surgery.

Ages: 1 Day to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 208 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2020-07-11 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is weight-adjusted cumulative morphine dose in the first 48 hours post-operatively. | 48 hours
  dose in micrograms per kilogram

SECONDARY OUTCOMES:
Incidence of adverse drug reactions | 96 hours
  1. Hemodynamic: hypotension or bradycardia, with the need for intervention by means of medication or a fluid bolus
  2. Decreased gastrointestinal motility or intestinal obstruction not directly related to the underlying diagnosis and not previously existing, with the need for intervention
  3. Vomiting
  4. Number of re-intubations (duration 48 hours)
  5. Pediatric delirium as measured by the Sophia Observation Withdrawal Symptoms scale Pediatric Delirium scale (SOS-PD, max score is 16/17, higher score more risk of pediatric delirium) or Cornell Assessment of Pediatric Delirium (CAPD, score > 9 gives increased risk of delirium) score.
Non-inferiority analysis of comparing the proportion of patients with one or more Numaric Rating Scale (NRS) scores of at least 4 between groups | 48 hours
  Numeric rating scale
The role of genetic polymorphisms in morphine metabolism | directly before surgery
  Genes involved in morphine metabolism: UGT2B7, ABCC3, and OCT1
Concomitant use of sedatives | 48 hours
  type and dose
mechanical ventilation duration in hours | immediately after surgery
The length of PICU stay | immediately after surgery
  Duration of PICU stay in both groups in days
Role of alarmins in the systemic inflammatory response (only at Wilhelmina Children's hospital) | 48 hours
  specific nuclear proteins to be determined (IL-1 alfa, IL-33, HMGB1)
Analysis of plasma morphine and paracetamo levels in relation to dose after cardia surgery using NONMEM (non-lineair mixed effects modelling). | 48 hours
  serum plasma levels of morphine and paracetamol

CONTACTS AND LOCATIONS:
Overall Officials: Enno Wildschut, MD, PhD, Principal Investigator — Erasmus Medical Center

IPD SHARING:
Plan to Share IPD: Yes
Study data can be shared with other researchers upon request.
Supporting Information: Study Protocol, SAP
Time Frame: not yet decided
Access Criteria: upon reasonable request

REFERENCES:
- [Derived] Zeilmaker-Roest G, de Vries-Rink C, van Rosmalen J, van Dijk M, de Wildt SN, Knibbe CAJ, Koomen E, Jansen NJG, Kneyber MCJ, Maebe S, Van den Berghe G, Haghedooren R, Vlasselaers D, Bogers AJJC, Tibboel D, Wildschut ED. Intermittent intravenous paracetamol versus continuous morphine in infants undergoing cardiothoracic surgery: a multi-center randomized controlled trial. Crit Care. 2024 Apr 30;28(1):143. doi: 10.1186/s13054-024-04905-3. PMID 38689310
- See also: published study protocol — https://pubmed.ncbi.nlm.nih.gov/29895289/